CLINICAL TRIAL: NCT05946525
Title: Ventilatory Variables in Subjects With Acute Respiratory Distress Syndrome Due to COVID-19
Status: Completed | Type: Observational
Sponsor: Hospital Donación Francisco Santojanni (Other)
Responsible Party: Principal Investigator, Marco Guillermo Bezzi, Licenciado Kinesiólogo Fisiatra, Hospital Donación Francisco Santojanni
Other Study IDs: HS9258
Record Dates: First submitted 2023-07-10; First posted 2023-07-14 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Respiratory Mechanics; Respiration, Artificial; Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Aspiration; Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Research question: Are the ventilatory variables related to mechanical power associated with the outcome of subjects who received mechanical ventilation (MV) for Acute Respiratory Distress Syndrome (ARDS) secondary to pneumonia (NMN) due to COVID-19?

DETAILED DESCRIPTION:
Primary Objective:

- To evaluate the association between the ventilatory variables of mechanical power and the outcome of the subjects in terms of mortality, days on MV and days free of MV at 28 days (both in survivors).

Secondary Objectives:

- Evaluate the association of demographic and gas exchange variables with the outcome of the subjects.

METHODOLOGY

Study design: retrospective and observational, analytical.

Operational definition of variables

Ventilatory variables:

* Global mechanical power: 0.098 × Tidal Volume × Respiratory Rate × (Peak Pressure - ½ Distension Pressure)
* Dynamic elastic mechanical power: 0.098 × Tidal Volume × Respiratory Rate × 0.5 × Distension Pressure
* Static elastic mechanical power: 0.098 × Tidal Volume × Respiratory Rate × PEEP
* Resistive mechanical power: 0.098 × Tidal Volume × Respiratory Rate × (Peak Pressure - Plateau Pressure)
* Cyclic Strain: DP x 4 + Respiratory Rate.
* Driving Pressure adjusted to predicted body weight: Driving Pressure / Tidal Volume (in ml / kg of predicted weight).

Demographic Variables:

* Age: in years.
* Sex: female / male.
* ARDS Classification:

  * Mild (PaO2 / FIO2 ≤ 300 mm Hg and > 200 mm Hg)
  * Moderate (PaO2 / FIO2 ≤ 200 mm Hg and > 100 mm Hg)
  * Severe (PaO2 / FIO2 ≤ 100 mm Hg)
* Body mass index: weight in kilograms divided by height in meters squared.

Gas Exchange Variables:

* Ventilatory quotient: (Respiratory Rate x Tidal Volume x PCO2) / (Predicted Weight x 100 ml x 37.5)
* Pa/FiO2: Arterial oxygen pressure/ Fraction of inspired oxygen Outcome Variables
* Mortality
* MV-free days at 28 days
* MV days Population and scope of study: Subjects registered in the ICU 2 database of the Francisco Santojanni Donation Hospital of the Autonomous City of Buenos Aires, who have received MV for ARDS with a confirmed diagnosis of COVID-19 pneumonia by polymerase chain reaction.

Study period: Data from subjects admitted from April 2020 to August 2021 will be analyzed.

Results analysis plan: A descriptive analysis of the clinical variables will be performed using the mean and standard deviation (SD), if the distribution is normal, or the median and interquartile range (IQR) otherwise.

Categorical variables will be presented as absolute number of presentation and percentage.

A value of p<0.05 will be considered as statistically significant.

SPSS software will be used for data analysis.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of pneumonia due to COVID-19.
* Need of mechanical ventilation in intensive care unit.

Exclusion Criteria:

* Patients with data loses

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admited to the intensive care unit with Mechanical ventilation due to ARDS with confirmed diagnosis of COVID-19 pneumonia by polymerase chain reaction (PCR),
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2023-02-10 (Actual); Primary Completion 2023-02-10 (Actual); Study Completion 2023-02-10 (Actual)

PRIMARY OUTCOMES:
global mechanical power | april 2020 to august 2021
  0,098 × Tidal Volume × Respiratory Rate × (Peak Pressure - ½ Driving Pressure)
Elastic Dynamic mechanical power | april 2020 to august 2021
  0,098 × Tidal Volume × Respiratory Rate × 0,5 × Driving Pressure
Elastic static mechanical power | april 2020 to august 2021
  0,098 × Tidal Volume × Respiratory Rate × PEEP
Resistive mechanical power | april 2020 to august 2021
  0,098 × Tidal Volume × Respiratory Rate × (Peak Pressure - Plateau Pressure)
Ciclic Strain | april 2020 to august 2021
  Driving Pressure x 4 + Respiratory Rate
Death | april 2020 to august 2021
  Death in intensive care unit
Suvival | april 2020 to august 2021
  discharge alive from intensive care unit

SECONDARY OUTCOMES:
ventilatory rate | april 2020 to august 2021
  (Respiratory Rate x Tidal Volume x PCO2) / (Predicted body weight x 100 ml x 37.5)
PaO2/FiO2 | april 2020 to august 2021
  partial pressure O2 divided O2 fraction

OTHER OUTCOMES:
age | april 2020 to august 2021
  age in years
sex | april 2020 to august 2021
  male or female
acute respiratory distress syndrome grade | april 2020 to august 2021
  severe (PaO2/FiO2 < 100) Moderate (PaO2/FiO2 100 to 200) and mild (PaO2/FiO2 > 200 to 300)
body mass index | april 2020 to august 2021
  body weight in kg divided squared heigh in m

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Santojanni, Buenos Aires, Argentina